CLINICAL TRIAL: NCT06235476
Title: Comparing the Effects of Three PROtein-enhancement Strategies on Exercise-induced Muscle Damage in Older Adults
Brief Title: Protein Intake and Exercise-induced Muscle Damage
Acronym: PROMO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Cosun (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 86007.091.23
Record Dates: First submitted 2023-12-21; First posted 2024-02-01 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-10

CONDITIONS: Sarcopenia
Keywords: Protein intake; Muscle damage; Nutritional intervention; Supplements; e-health
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Intervention Model Description: 4-arm intervention study
Who Masked: Participant, Investigator
Masking Description: The study consists of 4 arms of which 3 arms that receive a supplement and 1 arm that will use an e-health application to enhance protein intake. The 3 supplement arms are double-blind. The e-health arm is not; since it is not possible to blind either the participants in this group neither the investigators.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- animal-based protein (WP) (Experimental): Supplements and control (MPP, WP, CON) will be consumed as a drink or in a recipe for five subsequent weeks (30 g/day); four weeks preload and one week during the Four Days Marches. With this amount, we aim to increase the protein intake from <1.0g/kg/bw/d to >1.2g/kg/bw/d. Participants are allowed to dissolve the powder in a liquid of choice: we will provide several examples to the participants during the instructions.
  Interventions: Dietary Supplement: whey protein supplement
- plant-based protein (MPP) (Experimental): Supplements and control (MPP, WP, CON) will be consumed as a drink or in a recipe for five subsequent weeks (30 g/day); four weeks preload and one week during the Four Days Marches. With this amount, we aim to increase the protein intake from <1.0g/kg/bw/d to >1.2g/kg/bw/d. Participants are allowed to dissolve the powder in a liquid of choice: we will provide several examples to the participants during the instructions.
  Interventions: Dietary Supplement: mixed plant-based protein supplement
- protein-rich food products (PFP) (Experimental): PFP will receive digitally supported dietary intake counselling, with a focus on the use of protein-enriched food products in order to increase protein intake up to >1.2 k/kg/bw/d.
  Interventions: Other: e-health application
- control (CON) (Active Comparator): Supplements and control (MPP, WP, CON) will be consumed as a drink or in a recipe for five subsequent weeks (30 g/day); four weeks preload and one week during the Four Days Marches. With this amount, we aim to increase the protein intake from <1.0g/kg/bw/d to >1.2g/kg/bw/d. Participants are allowed to dissolve the powder in a liquid of choice: we will provide several examples to the participants during the instructions.
  Interventions: Dietary Supplement: isocaloric carbohydrate control

INTERVENTIONS:
Dietary Supplement: whey protein supplement — Daily dosage of the supplements will be 30 gram, preferably consumed in the morning and post-exercise or prior to sleep.
  Arms: animal-based protein (WP)
Dietary Supplement: mixed plant-based protein supplement — Daily dosage of the supplements will be 30 gram, preferably consumed in the morning and post-exercise or prior to sleep.
  Arms: plant-based protein (MPP)
Other: e-health application — Daily use of an e-health application with dietary intake counselling to increase protein intake. The overall goal of these advices is to increase protein intake from <1.0g/kg/bw/d to >1.2g/kg/bw/d which is approximately 30 grams of additional protein per day (similar to the other arms of the intervention).
  Arms: protein-rich food products (PFP)
Dietary Supplement: isocaloric carbohydrate control — Daily dosage of the supplements will be 30 gram, preferably consumed in the morning and post-exercise or prior to sleep.
  Arms: control (CON)

SUMMARY:
The goal of this clinical trial is to test the effect of different protein-enhancement strategies versus carbohydrate control on exercise-induced muscle damage in physically active older adults. The main question it aims to answer is:

What is the effect of three different protein-enhancement strategies (whey protein (WP), mixed plant-based protein (MPP), and use of protein-rich food products (PFP) on exercise-induced muscle damage in older adults compared to isocaloric carbohydrate control?

Participants will:

* Use a protein-enhancement strategy (WP, MPP or PFP) or carbohydrate control for a total of 5 weeks;
* Participate in a single walking bound (30/40/50 km) two weeks after the start of the study;
* Participate in a consecutive walking bound (4 days of 30/40/50 km) in the last week of the study period;
* Complete different questionnaires and give blood samples to test for muscle damage.

ELIGIBILITY:
Inclusion Criteria:

* 60 years or older
* Registered for the Nijmegen Four Days Marches (i.e., able to walk 30-50 km/day)
* A habitual protein intake <1.0 g/kg/d based on the protein 55+ (PRO55+) screening tool
* Able to understand and perform the study procedures
* Able to use a mobile device

Exclusion Criteria:

* Allergic or sensitive for milk proteins, or lactose intolerant
* Diagnosed type I or type II diabetes mellitus
* Diagnosed intestinal diseases influencing the uptake of protein (i.e., active inflammatory bowel disease, Crohn's disease)
* Consumption of other freely available protein supplements during the study period.
* If the subject intends to perform additional exercise bouts that cause muscle damage in the 4 days before the single- and multiple exercise bouts.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 199 (Actual)
Dates: Start 2024-06-10 (Actual); Primary Completion 2024-07-19 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
serum creatine kinase (CK) levels | Measured 8 times in total. Once pre-single exercise, two times post-single exercise (within 2h after and around 24h after) and 2 weeks later: once pre-multiple day exercise and four times post-multiple day exercise (within 2h post-exercise)
  Exercise-induced muscle damage. Non-fasted venous blood samples will be drawn from the antecubital vein at each pre-exercise and post-exercise visit. Based on previous research it is expected that time-dependent exercise-induced increase in creatine kinase (CK) levels are significantly different between protein groups and control, but not within protein groups. Multiple peak post-exercise CK concentrations (several hours to up to 48h post exercise) will be compared to pre-exercise CK levels to compare the effect of different protein enhancing strategies versus carbohydrate control.

SECONDARY OUTCOMES:
serum lactate dehydrogenase (LDH) levels | Measured 8 times in total. Once pre-single exercise, two times post-single exercise (within 2h after and around 24h after) and 2 weeks later: once pre-multiple day exercise and four times post-multiple day exercise (within 2h post-exercise)
  (Muscle) cell damage. Non-fasted venous blood samples will be drawn from the antecubital vein at each pre-exercise and post-exercise visit.
muscle soreness | Measured 8 times in total. Once pre-single exercise, two times post-single exercise (within 2h after and around 24h after) and 2 weeks later: once pre-multiple day exercise and four times post-multiple day exercise (within 2h post-exercise)
  Muscle soreness is measured via the the Numeric Pain Scale (from 0 to 10, a higher score means more muscle soreness.
muscle function | Measured 8 times in total. Once pre-single exercise, two times post-single exercise (within 2h after and around 24h after) and 2 weeks later: once pre-multiple day exercise and four times post-multiple day exercise (within 2h post-exercise)
  Maximal handgrip strength is measured to the nearest 0.5 kg using a hand dynamometer. The participants is seated in a chair with the shoulders adducted and neutrally rotated and elbow flexed at 90o. Three consecutive measurements of handgrip strength will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Hopman, prof. dr., Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboudumc, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Individual Participant Data (IPD) will be shared with researchers within the department of Medical Biosciences of the Radboud University Medical Center (Radboudumc). The department has a database of data from the past 15 years of Four Day Marches data. This research data will be added to the database. Data may be shared with other researchers upon request.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data will become available after completion of the study and will be available for at least 15 years.
Access Criteria: IPD will be shared with researchers within the department of Medical Biosciences of the Radboudumc. Data may be shared with other researchers upon request.